CLINICAL TRIAL: NCT02637739
Title: Office Hysteroscopy as a Diagnostic Tool of Pregnancy of Unknown Location
Brief Title: Hysteroscopy for Pregnancy of Unknown Location
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hung Lin, M.D., Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SKH-8302-104_DR-18
Record Dates: First submitted 2015-12-06; First posted 2015-12-22 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Pregnancy
Keywords: hysteroscope
MeSH Terms: interventions — Hysteroscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pregnancy of unknown location (Experimental): pregnant women of at least 5 weeks by last menstrual period and transvaginal ultrasound did not revealed intra-uterine pregnancy or ectopic pregnancy Intervention: hysteroscope
  Interventions: Device: hysteroscope

INTERVENTIONS:
Device: hysteroscope — Women of PUL with β-hCG > 1000 IU/L or abnormal β-hCG trend (increase < 66% or decrease < 15%) were offered HSC.

SUMMARY:
About 10% of early pregnancies can not be visualized by transvaginal ultrasound (TVU) on first visit and are classified as pregnancy of unknown location (PUL). The etiology includes ongoing intra-uterine pregnancy, failing pregnancy, or ectopic pregnancy. Early diagnosis of ectopic pregnancy is important because it allows conservative treatment. Serum β-hCG, D&C, and laparoscopy are routinely used as diagnostic methods. The purpose of the study is to evaluate if the less invasive office hysteroscopy (HSC) can help diagnose PUL.

DETAILED DESCRIPTION:
If TVU showed no evidence of intra-uterine and extra-uterine pregnancy, a blood test for β-hCG was done. If β-hCG was < 1000 IU/L, the woman was followed with β-hCG 2 days later. Women with β-hCG > 1000 IU/L or abnormal β-hCG trend (increase < 66% or decrease < 15%) were offered HSC. If gestational tissues were visualized, ectopic pregnancy was ruled out. Otherwise, the tentative diagnosis was ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women with PUL

Exclusion Criteria:

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
percentage of women with PUL waived from laparoscopic examination | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gong-Jhe Wu, Study Director — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Shin-Kong Wu-Ho-Su Memerial Hospital, Taipei, Taiwan